CLINICAL TRIAL: NCT01185951
Title: TENDOSHOCK-2010 - Combined Sclerosing Therapy, Extracorporeal Shockwave Therapy, Eccentric Training and Topical Glyceryl Trinitrate for Athletic Tendinopathies
Brief Title: TENDOSHOCK-2010 Combination Therapy for Athletic Tendinopathies
Acronym: TENDOSHOCK
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: PD Dr. Karsten Knobloch, Plastic, Hand and Reconstructive Surgery, Hannover Medical School, Germany
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TENDOSHOCK-2010
Record Dates: First submitted 2010-08-17; First posted 2010-08-20 (Estimated); Last update posted 2010-08-20 (Estimated); Status verified 2010-08

CONDITIONS: Tendinopathy; Epicondylitis
Keywords: Achilles Tendon; Patella; Allergy; Necrosis; Infection
MeSH Terms: conditions — Tendinopathy; Patella Fracture; Hypersensitivity; Necrosis; Infections | interventions — Polidocanol; Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Achilles tendinopathy (Active Comparator): Patients suffering both, insertional and midportion Achilles tendinopathy seeking medical help. All patients were evaluated with a standardized Power-Doppler ultrasound to detect the level of neovascularisation at the point of pain.
  Interventions: Drug: Polidocanol; Device: Focused extracorporeal shock wave therapy; Drug: Topical NO; Behavioral: Painful eccentric training in Achilles tendinopathy
- Patella tendinopathy (Active Comparator): Patients suffering patella tendinopathy seeking medical help. All patients were evaluated with a standardized Power-Doppler ultrasound to detect the level of neovascularisation at the point of pain.
  Interventions: Drug: Polidocanol; Device: Focused extracorporeal shock wave therapy; Drug: Topical NO; Behavioral: Painful eccentric training for patella tendinopathy on 25° decline board
- Epikondylitis (Active Comparator): Patients suffering both, lateral (tennis elbow) or medial (golfers' elbow) elbow tendinopathy seeking medical help. All patients were evaluated with a standardized Power-Doppler ultrasound to detect the level of neovascularisation at the point of pain.
  Interventions: Drug: Polidocanol; Device: Focused extracorporeal shock wave therapy; Drug: Topical NO; Behavioral: Painful eccentric training for elbow tendinopathy using Thera-Band Flex-Bar

INTERVENTIONS:
Drug: Polidocanol — Power-Doppler-guided extratendinous sclerosing therapy using Polidocanol 0.5% up to 2ml every 6-8 weeks
Device: Focused extracorporeal shock wave therapy — Focused extracorporeal shock wave therapy using a STORZ Duolith machine 2000 Impulses 0.25mJ/mm2 every 6-8 weeks
Drug: Topical NO — Topical nitroglycerine (Nitrolingualspray(R)) 2x2 hubs per day over 6 months daily on the painful tendon
Behavioral: Painful eccentric training in Achilles tendinopathy — Painful eccentric training for Achilles tendinopathy on a stair single-stance with 6x15 repetitions per leg and day over at least 12 weeks
  Arms: Achilles tendinopathy
Behavioral: Painful eccentric training for patella tendinopathy on 25° decline board — Painful eccentric training for patella tendinopathy on a 25° decline board single-stance with 6x15 repetitions per leg and day over at least 12 weeks
  Arms: Patella tendinopathy
Behavioral: Painful eccentric training for elbow tendinopathy using Thera-Band Flex-Bar — Painful eccentric training for elbow tendinopathy using a green coloured Thera-Band Flex-Bar with painful supination and pronation with 6x15 repetitions per day over at least 12 weeks
  Arms: Epikondylitis

SUMMARY:
Athletic tendinopathies of the upper and lower extremity are often therapeutically challenging. Colour and Power-Doppler-ultrasound visualizes pathological neovessels in painful tendons, which are associated with pain-mediating nerve fibres in such tendinopathies. These neovessels are represented by an increased capillary blood flow at the point of pain. Painful eccentric training reduces pain and improves function in Achilles tendinopathy substantially (evidence level Ib). Shock wave therapy in combination with eccentric training is superior to eccentric training alone (evidence level Ib). Long-term results suggest a collagen induction and reduced pain following topical glyceryl trinitrate (NO) (evidence level Ib). Colour- and Power-Doppler-guided sclerosing therapy using polidocanol reduces pain, improves function and may lead to tendon remodelling (evidence level Ib). Pain-restricted sport beyond pain level 5/10 during therapy is recommended (evidence level Ib). 3x10min of cryotherapy reduce pain and capillary blood flow (evidence level Ib). The role of proprioceptive training in tendinopathy has to be determined in future randomized-controlled trials (evidence level II).

The investigators thought to evaluate the combination of the aforementioned individually successfully therapeutic options in athletes to shorten the recovery period and return to play interval.

DETAILED DESCRIPTION:
Interventions:

Combined Power-Doppler-guided sclerosing therapy using Polidocanol (0.5%, 2ml) in 6-8 week intervals combined with extracorporeal focused shockwave therapy (STORZ Duolith 2000impulses 0.25mJ/mm2) every 6-8weeks plus painful daily eccentric training plus daily topical NO

ELIGIBILITY:
Inclusion Criteria:

* Painful tendons at the Achilles tendon (both insertional and mid-portion tendinopathy)
* patella tendinopathy
* elbow tendinopathy
* informed consent

Exclusion Criteria:

* no informed consent
* no painful tendons
* allergy against Polidocanol
* current treatment with Marcumar

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2007-01; Primary Completion 2010-08 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Functional impairment of the Achilles tendon using VISA-A score [0=worse, 100=perfect] | up to 4 years
  Score of patient-related outcome measure: Achilles tendon: VISA-A [0=worse, 100=perfect] derived from eight validated questions on pain and function during activities of daily living
Functional impairment of the patella tendon according to the VISA-P score [0=worse, 100=perfect] | up to 4 years
  Score of patient-related outcome measure: Patella tendon: VISA-P [0=worse, 100=perfect] derived from eight validated questions on pain and function during daily activities
Functional impairment due to epicondylitis measured by the DASH score [0=perfect, 100=worse] | up to four years
  Score of patient-related outcome measure: Epicondylitis: DASH score [0=perfect, 100=worse] derived from 30 validated questions regarding the impairment in activities of daily living

SECONDARY OUTCOMES:
Pain level at rest [VAS 0-10] | up to 4 years
Pain level at exertion [VAS 0-10] | up to 4 years
Patient satisfaction on Likert scale [1-6] | up to 4 years
  Patient satisfaction on Likert scale from 1=perfect, wholy satisfied, to 6=worst, dissatisfied

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Knobloch, MD, Principal Investigator — Hannover Medical School, Germany
Locations (1):
- Hannover Medical School, Plastic, Hand and Reconstructive Surgery, Hanover, Germany

REFERENCES:
- [Background] Knobloch K, Schreibmueller L, Kraemer R, Jagodzinski M, Vogt PM, Redeker J. Gender and eccentric training in Achilles mid-portion tendinopathy. Knee Surg Sports Traumatol Arthrosc. 2010 May;18(5):648-55. doi: 10.1007/s00167-009-1006-7. Epub 2009 Dec 9. PMID 19997901
- [Background] Osadnik R, Redeker J, Kraemer R, Vogt PM, Knobloch K. Microcirculatory effects of topical glyceryl trinitrate on the Achilles tendon microcirculation in patients with previous Achilles tendon rupture. Knee Surg Sports Traumatol Arthrosc. 2010 Jul;18(7):977-81. doi: 10.1007/s00167-009-0958-y. Epub 2009 Oct 31. PMID 19882141
- [Background] Kraemer R, Knobloch K. A soccer-specific balance training program for hamstring muscle and patellar and achilles tendon injuries: an intervention study in premier league female soccer. Am J Sports Med. 2009 Jul;37(7):1384-93. doi: 10.1177/0363546509333012. PMID 19567665
- [Background] Knobloch K. Sclerosing polidocanol injections in Achilles tendinopathy in high level athletes. Knee Surg Sports Traumatol Arthrosc. 2008 Nov;16(11):1061-2; author reply 1063. doi: 10.1007/s00167-008-0613-z. Epub 2008 Sep 13. No abstract available. PMID 18791700
- [Background] Knobloch K, Yoon U, Vogt PM. Acute and overuse injuries correlated to hours of training in master running athletes. Foot Ankle Int. 2008 Jul;29(7):671-6. doi: 10.3113/FAI.2008.0671. PMID 18785416
- [Background] Knobloch K, Schreibmueller L, Longo UG, Vogt PM. Eccentric exercises for the management of tendinopathy of the main body of the Achilles tendon with or without an AirHeel Brace. A randomized controlled trial. B: Effects of compliance. Disabil Rehabil. 2008;30(20-22):1692-6. doi: 10.1080/09638280701785676. PMID 18720130
- [Background] Knobloch K, Schreibmueller L, Longo UG, Vogt PM. Eccentric exercises for the management of tendinopathy of the main body of the Achilles tendon with or without the AirHeel Brace. A randomized controlled trial. A: effects on pain and microcirculation. Disabil Rehabil. 2008;30(20-22):1685-91. doi: 10.1080/09638280701786658. PMID 18720121
- [Background] Knobloch K, Thermann H. [Achilles tendinopathy--modern evidence-based recommendations]. MMW Fortschr Med. 2008 Jun 26;150(26-27):46-9; quiz 50. No abstract available. German. PMID 18681232
- [Background] Knobloch K, Grasemann R, Spies M, Vogt PM. Midportion achilles tendon microcirculation after intermittent combined cryotherapy and compression compared with cryotherapy alone: a randomized trial. Am J Sports Med. 2008 Nov;36(11):2128-38. doi: 10.1177/0363546508319313. Epub 2008 Jul 18. PMID 18641371
- [Background] Knobloch K. The role of tendon microcirculation in Achilles and patellar tendinopathy. J Orthop Surg Res. 2008 Apr 30;3:18. doi: 10.1186/1749-799X-3-18. PMID 18447938
- [Background] Knobloch K, Schreibmueller L, Meller R, Busch KH, Spies M, Vogt PM. Superior Achilles tendon microcirculation in tendinopathy among symptomatic female versus male patients. Am J Sports Med. 2008 Mar;36(3):509-14. doi: 10.1177/0363546507309313. Epub 2007 Oct 30. PMID 17971505
- [Background] Knobloch K, Kraemer R, Jagodzinski M, Zeichen J, Meller R, Vogt PM. Eccentric training decreases paratendon capillary blood flow and preserves paratendon oxygen saturation in chronic achilles tendinopathy. J Orthop Sports Phys Ther. 2007 May;37(5):269-76. doi: 10.2519/jospt.2007.2296. PMID 17549956
- [Background] Knobloch K, Spies M, Busch KH, Vogt PM. Sclerosing therapy and eccentric training in flexor carpi radialis tendinopathy in a tennis player. Br J Sports Med. 2007 Dec;41(12):920-1. doi: 10.1136/bjsm.2007.036558. Epub 2007 May 11. PMID 17496066
- [Background] Knobloch K, Thermann H, Hufner T. [Achilles tendon rupture--early functional and surgical options with special emphasis on rehabilitation issues]. Sportverletz Sportschaden. 2007 Mar;21(1):34-40. doi: 10.1055/s-2007-963040. German. PMID 17385103
- [Background] Knobloch K, Grasemann R, Spies M, Vogt PM. Intermittent KoldBlue cryotherapy of 3x10 min changes mid-portion Achilles tendon microcirculation. Br J Sports Med. 2007 Jun;41(6):e4. doi: 10.1136/bjsm.2006.030957. Epub 2006 Nov 30. PMID 17138636
- [Background] Knobloch K. Eccentric training in Achilles tendinopathy: is it harmful to tendon microcirculation? Br J Sports Med. 2007 Jun;41(6):e2; discussion e2. doi: 10.1136/bjsm.2006.030437. Epub 2006 Nov 24. PMID 17127721
- [Background] Knobloch K, Grasemann R, Jagodzinski M, Richter M, Zeichen J, Krettek C. Changes of Achilles midportion tendon microcirculation after repetitive simultaneous cryotherapy and compression using a Cryo/Cuff. Am J Sports Med. 2006 Dec;34(12):1953-9. doi: 10.1177/0363546506293701. Epub 2006 Sep 22. PMID 16998082